CLINICAL TRIAL: NCT03019393
Title: Effect of Red Meat Intake on Occurrence of Serum Non-transferrin Bound Iron (NTBI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Walczyk (Other)
Responsible Party: Sponsor-Investigator, Thomas Walczyk, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-441
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: non-transferrin bound iron (NTBI); Red meat; Non-transferrin bound iron (NTBI) in serum
MeSH Terms: interventions — Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Beef (Other): Beef topside fully cooked, 200g
  Interventions: Other: Beef

INTERVENTIONS:
Other: Beef — 200 g beef topside which is fully cooked will be provided to participant after overnight fast. The intervention is one time only.

SUMMARY:
This study aims to evaluate the effect of red meat intake on occurrence of non-transferrin bound iron (NTBI)

DETAILED DESCRIPTION:
During Visit 1, blood samples will be collected to assess iron status. During Visit 2, after an overnight fast, participant will be given a standardized meal (rice and potatoes) with a portion of cooked beef (200 g). Blood samples will be collected right before and 2 hour after the meal for NTBI analysis.

NTBI concentration before and after meal consumption will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy male volunteers (21 - 45 years old)
* C-reactive protein (CRP) < 5 mg/L

Exclusion Criteria:

* Blood donation or significant blood loss (e.g. surgery) within the past 4 months
* Regular intake of iron and other nutrient supplements within the past 4 months
* Regular intake of medication except oral contraceptives
* Acute or recent inflammatory or infectious symptoms
* Chronic gastrointestinal disorders or metabolic diseases
* Smoking
* Coeliac disease or gluten-related disorders
* Iron deficiency anemia (Hb < 14 g/dL for males) with serum ferritin concentration < 30 ng/mL)
* Non-iron deficiency anemia (serum ferritin concentration within normal range (30 - 300 ng/mL for males) but low hemoglobin (< 14 g/dL for males)
* Iron overload conditions (serum ferritin concentration > 300 ng/mL for males)
* Known hereditary disorders of iron metabolism

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serum non-transferrin bound iron (NTBI) after consumption of red meat | 2 hour post meal administration
  Blood samples collected 2 h after consumption of red meat will be analyzed for non-transferrin bound iron (NTBI) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walczyk, Ph.D, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore; National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trumbo P, Yates AA, Schlicker S, Poos M. Dietary reference intakes: vitamin A, vitamin K, arsenic, boron, chromium, copper, iodine, iron, manganese, molybdenum, nickel, silicon, vanadium, and zinc. J Am Diet Assoc. 2001 Mar;101(3):294-301. doi: 10.1016/S0002-8223(01)00078-5. No abstract available. PMID 11269606
- [Background] Monsen ER, Hallberg L, Layrisse M, Hegsted DM, Cook JD, Mertz W, Finch CA. Estimation of available dietary iron. Am J Clin Nutr. 1978 Jan;31(1):134-41. doi: 10.1093/ajcn/31.1.134. PMID 619599
- [Background] Papanikolaou G, Pantopoulos K. Iron metabolism and toxicity. Toxicol Appl Pharmacol. 2005 Jan 15;202(2):199-211. doi: 10.1016/j.taap.2004.06.021. PMID 15629195
- [Background] Hutchinson C, Al-Ashgar W, Liu DY, Hider RC, Powell JJ, Geissler CA. Oral ferrous sulphate leads to a marked increase in pro-oxidant nontransferrin-bound iron. Eur J Clin Invest. 2004 Nov;34(11):782-4. doi: 10.1111/j.1365-2362.2004.01416.x. No abstract available. PMID 15530152
- [Background] Schumann K, Kroll S, Romero-Abal ME, Georgiou NA, Marx JJ, Weiss G, Solomons NW. Impact of oral iron challenges on circulating non-transferrin-bound iron in healthy Guatemalan males. Ann Nutr Metab. 2012;60(2):98-107. doi: 10.1159/000336177. Epub 2012 Mar 6. PMID 22398912